CLINICAL TRIAL: NCT00457392
Title: A Multicenter, Randomized, Double-Blind, Controlled Phase 3, Efficacy And Safety Study Of Sunitinib (SU011248) In Patients With Advanced/Metastatic Non-Small Cell Lung Cancer Treated With Erlotinib
Brief Title: A Study In Patients With Non-Small Cell Lung Cancer To Test If Erlotinib Plus SU011248 Is Better Than Erlotinib Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A6181087; SUN1087
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Non-small cell lung cancer; sunitinib; erlotinib; Phase 3
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: erlotinib; Drug: sunitinib
- 2 (Active Comparator)
  Interventions: Drug: erlotinib; Drug: placebo

INTERVENTIONS:
Drug: erlotinib — plus erlotinib 150 mg daily by tablets in a continuous regimen until progression or unacceptable toxicity
  Arms: 1
Drug: sunitinib — Sunitinib 37.5 mg daily by oral capsules in a continuous regimen
  Arms: 1
Drug: erlotinib — plus erlotinib 150 mg daily by tablets in a continuous regimen until progression or unacceptable toxicity
  Arms: 2
Drug: placebo — Placebo daily by oral capsules in a continuous regimen
  Arms: 2

SUMMARY:
This study will test whether treatment with erlotinib plus SU011248 is better than erlotinib alone in patients with advanced/metastatic lung cancer who have received previous treatment with a platinum-based regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced/metastatic non-small cell lung cancer
* Prior treatment with no more than 2 chemotherapy regimens including a platinum-based regimen

Exclusion Criteria:

* Prior treatment with any receptor tyrosine kinase inhibitors, VEGF inhibitor (with the exception of bevacizumab) or other angiogenesis inhibitors
* History of or known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (182):
- United States (56):
  - Pfizer Investigational Site, Florence, Alabama
  - Pfizer Investigational Site, Muscle Shoals, Alabama
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Antioch, California
  - Pfizer Investigational Site, Burbank, California
  - Pfizer Investigational Site, Downey, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Montebello, California
  - Pfizer Investigational Site, Pleasant Hill, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Leandro, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Fairfield, Connecticut
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Cocoa Beach, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Merritt Island, Florida
  - Pfizer Investigational Site, Rockledge, Florida
  - Pfizer Investigational Site, Titusville, Florida
  - Pfizer Investigational Site, Athens, Georgia
  - Pfizer Investigational Site, Aurora, Illinois
  - Pfizer Investigational Site, Goshen, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Council Bluffs, Iowa
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Lafayette, Louisiana
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Columbus, Mississippi
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Jamaica, New York
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Grapevine, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Bountiful, Utah
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Provo, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Sandy City, Utah
  - Pfizer Investigational Site, West Valley City, Utah
  - Pfizer Investigational Site, Kennewick, Washington
- Argentina (3):
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires F.D.
  - Pfizer Investigational Site, Córdoba, Córdoba Province
  - Pfizer Investigational Site, Buenos Aires
- Austria (3):
  - Pfizer Investigational Site, Grimmenstein
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Linz
- Belgium (3):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
- Brazil (4):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Barretos, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (8):
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, Lévis, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Rimouski, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Chile (3):
  - Pfizer Investigational Site, Santiago, Chile
  - Pfizer Investigational Site, Independencia, Santiago, RM
  - Pfizer Investigational Site, Providencia, Santiago, RM
- Pfizer Investigational Site, Medellín, Antioquia, Colombia
- Czechia (8):
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Nová Ves pod Pleší
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Ostrava-Poruba
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Pribram V
  - Pfizer Investigational Site, Tábor
  - Pfizer Investigational Site, Ústí nad Labem
- Denmark (4):
  - Pfizer Investigational Site, Herlev
  - Pfizer Investigational Site, Hilleroed
  - Pfizer Investigational Site, Koebenhavn OE
  - Pfizer Investigational Site, Odense
- Germany (13):
  - Pfizer Investigational Site, Bad Berka
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Ebensfeld
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Gauting
  - Pfizer Investigational Site, Großhansdorf
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Homburg
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Tübingen
  - Pfizer Investigational Site, Wiesbaden
- Greece (4):
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Alexandroupoli
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Kifisia, Athens
- Hong Kong (3):
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Shatin, NT
  - Pfizer Investigational Site, Tuenmen
- Hungary (6):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Deszk
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Mátraháza
  - Pfizer Investigational Site, Székesfehérvár
  - Pfizer Investigational Site, Zalaegerszeg-Pozva
- Italy (10):
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Grosseto
  - Pfizer Investigational Site, Mantova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Monza (MI)
  - Pfizer Investigational Site, Novara
  - Pfizer Investigational Site, Orbassano (TO)
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Rozzano (MI)
- Netherlands (7):
  - Pfizer Investigational Site, Enschede, Overijssel
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Arnhem
  - Pfizer Investigational Site, Harderwijk
  - Pfizer Investigational Site, Maastricht
  - Pfizer Investigational Site, Rotterdam
- Norway (5):
  - Pfizer Investigational Site, Kristiansand
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Stavanger
  - Pfizer Investigational Site, Tromsø
  - Pfizer Investigational Site, Trondheim
- Poland (5):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Opole
  - Pfizer Investigational Site, Otwock
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Zielona Góra
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Slovakia (5):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Kvetnica Pri Poprade
  - Pfizer Investigational Site, Nitra-Zobor
  - Pfizer Investigational Site, Žilina
- Pfizer Investigational Site, Seoul, South Korea
- Spain (10):
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, A Coruña, La Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Pfizer Investigational Site, Dos Hermanas, Sevilla
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
- Pfizer Investigational Site, Genolier, Switzerland
- Taiwan (3):
  - Pfizer Investigational Site, Gwei Shan Township, Taoyuan County
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
- Thailand (3):
  - Pfizer Investigational Site, Pathumwan, Bangkok
  - Pfizer Investigational Site, Amphoe Mueang, Chiang Mai
  - Pfizer Investigational Site, Bangkok
- United Kingdom (11):
  - Pfizer Investigational Site, Bebington, Wirral
  - Pfizer Investigational Site, Cambridge
  - Pfizer Investigational Site, Derby
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Keighley, West Yorkshire
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Peterborough
  - Pfizer Investigational Site, Rhyl, Denbigshire
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Southampton
  - Pfizer Investigational Site, Yeovil, Somerset

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181087&StudyName=A%20Study%20In%20Patients%20With%20Non-Small%20Cell%20Lung%20Cancer%20To%20Test%20If%20Erlotinib%20Plus%20SU011248%20Is%20Better%20Than%20Erlotinib%20Alone

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib + Erlotinib: Sunitinib capsule administered orally at a dose of 37.5 milligram (mg) daily (continuous regimen) in a 4 week cycle. Erlotinib administered orally at a dose of 150 mg daily.
- Erlotinib: Placebo capsule matched to sunitinib administered orally daily (continuous regimen) in a 4 week cycle. Erlotinib 150 mg tablet orally daily.
Period: Overall Study
Arm/Group | Sunitinib + Erlotinib | Erlotinib
Started | 480 | 480
Treated | 473 | 477
Completed | 0 | 0
Not Completed | 480 | 480
Not completed — Objective Progression or Relapse | 229 | 296
Not completed — Death | 106 | 106
Not completed — Adverse Event | 84 | 41
Not completed — Global Deterioration of Health Status | 22 | 8
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Lost to Follow-up | 6 | 7
Not completed — Protocol Violation | 4 | 3
Not completed — Other | 7 | 4
Not completed — Study Terminated by Sponsor | 1 | 4
Not completed — Randomized, Not Treated | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib + Erlotinib | Erlotinib | Total
Number analyzed (Participants) | 480 | 480 | 960
Age Continuous [Mean (Standard Deviation); unit: Years] | 61.10 (9.97) | 60.80 (9.13) | 60.90 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 196 | 379
  Male | 297 | 284 | 581

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is the duration from assignment to study medication to death. For participants who are alive, overall survival is censored at the last contact.
Time Frame: Baseline to death or 28 days after last dose for the last participant
Population: The Full Analysis (FA) set included all participants who were randomized, with study drug assignment designated according to actual randomization, regardless of whether participants received study drug according to the randomization schedule, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib + Erlotinib | Erlotinib
Number analyzed (Participants) | 480 | 480
Months | 9.0 [8.4 to 10.2] | 8.5 [7.4 to 9.8]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib; Differences in OS between treatment arms was analyzed by the 1-sided log rank test, stratified for smoking status (ever versus never), prior bevacizumab therapy (yes versus no) and epidermal growth factor receptor (EGFR) status (positive, versus negative, versus unknown); Test type: Superiority or Other; p = 0.1933, Log Rank — p-value was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.942, 95% CI 2-sided [0.822 to 1.079]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time in weeks from assignment to study medication to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline to disease progression or death due to any cause or 28 days after last dose
Population: The FA set included all participants who were randomized, with study drug assignment designated according to actual randomization, regardless of whether participants received study drug according to the randomization schedule, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib
Number analyzed (Participants) | 480 | 480
Weeks | 15.5 [13.1 to 16.1] | 8.7 [8.3 to 12.8]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib; Differences in PFS between treatment arms was analyzed by the 1-sided log rank test, stratified for smoking status (ever versus never), prior bevacizumab therapy (yes versus no) and EGFR status (positive, versus negative, versus unknown); Test type: Superiority or Other; p = 0.0023, Log Rank — No p-value is adjusted for multiple comparisons for PFS; One-sided log-rank test with alpha=0.025 was used; Hazard Ratio (HR) = 0.807, 95% CI 2-sided [0.695 to 0.937]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.0. Confirmed response are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as disappearance of all lesions (target and/or non target). PR are those with at least 30% decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: Baseline to disease progression or discontinuation from study or 28 days after last dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib
Number analyzed (Participants) | 480 | 480
Percentage of participants | 10.60 [8.01 to 13.73] | 6.90 [4.78 to 9.52]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib; The Cochran-Mantel-Haenszel (CMH) test stratified for smoking status (ever versus never), prior bevacizumab therapy (yes versus no) and EGFR status (positive, versus negative, versus unknown) was used to compare ORR between the 2 treatment arms. The relative risk ratio estimator was used to contrast the treatment effects on response rates. A point estimate of relative risk ratio and 2-sided 95% CI was calculated; Test type: Superiority or Other; p = 0.0471, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.514, 95% CI 2-sided [1.002 to 2.289]

4. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7.
Time Frame: Baseline to disease progression or death or discontinuation from study or 28 days after last dose
Population: DR was calculated for the subgroup of participants from the FA set, with a confirmed objective tumor response.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib
Number analyzed (Participants) | 51 | 33
Weeks | 39.6 [31.3 to 48.9] | 32.3 [24.2 to 48.0]

5. Secondary Outcome: One-year Survival Probability
Description: The 1 year survival probability was defined as the probability of survival at one year after the date of the start of the study treatment based on the Kaplan Meier estimate.
Time Frame: Baseline until death or until 28 days after last dose for the last participant
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent chance of survival
Arm/Group | Sunitinib + Erlotinib | Erlotinib
Number analyzed (Participants) | 480 | 480
Percent chance of survival | 40.0 [35.4 to 44.2] | 37.0 [32.8 to 41.6]

6. Secondary Outcome: EuroQol 5-Dimension Questionnaire (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in total score range -0.594 to 1.000; higher score indicates better health state.
Time Frame: Baseline and End of Treatment (EOT) or Withdrawal
Population: Patients Reported Outcome (PRO) Analysis Set included participants from the FA population who had at least one EQ-5D assessment while on treatment. The 'n' signifies those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sunitinib + Erlotinib | Erlotinib
Number analyzed (Participants) | 451 | 465
Units on a scale
  Baseline | 0.750 (0.239) | 0.716 (0.263)
  End of Treatment (n= 285, 301) | 0.615 (0.348) | 0.598 (0.339)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib + Erlotinib | Erlotinib
Serious Adverse Events (participants affected / at risk) | 207/473 | 181/477
Other Adverse Events (participants affected / at risk) | 463/473 | 461/477
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Erlotinib (N=473) | Erlotinib (N=477)
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 0
Pericardial effusion (Cardiac disorders) | 3 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 22 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 5
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 11 | 8
Asthenia (General disorders) | 11 | 4
Chest pain (General disorders) | 0 | 4
Death (General disorders) | 2 | 4
Disease progression (General disorders) | 70 | 61
Euthanasia (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 1
General physical health deterioration (General disorders) | 6 | 3
Irritability (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 6 | 4
Sudden death (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 2 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 7 | 13
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pyonephrosis (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Body temperature increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 9 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Meningorrhagia (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 1
Paralysis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Aggression (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Sopor (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 2
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Erlotinib (N=473) | Erlotinib (N=477)
Anaemia (Blood and lymphatic system disorders) | 51 | 23
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 20 | 3
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 9 | 1
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 34 | 4
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 32 | 2
Angina pectoris (Cardiac disorders) | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 4
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 0
Extrasystoles (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 3 | 0
Palpitations (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 5 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 3 | 6
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 3
Trichomegaly (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Dysacusis (Ear and labyrinth disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 2
Ear pruritus (Ear and labyrinth disorders) | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 6 | 9
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Adrenal disorder (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 2 | 2
Parathyroid haemorrhage (Endocrine disorders) | 0 | 1
Blepharitis (Eye disorders) | 1 | 2
Cataract (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 2
Conjunctivitis (Eye disorders) | 19 | 20
Conjunctivitis allergic (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 7 | 9
Erythema of eyelid (Eye disorders) | 0 | 1
Eye allergy (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 1
Eye irritation (Eye disorders) | 2 | 3
Eye oedema (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 0 | 2
Eye pruritus (Eye disorders) | 3 | 4
Eyelid disorder (Eye disorders) | 0 | 1
Eyelid function disorder (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 6 | 1
Eyelid pain (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 3 | 0
Keratoconjunctivitis sicca (Eye disorders) | 2 | 0
Lacrimal gland enlargement (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 8 | 3
Lenticular opacities (Eye disorders) | 0 | 1
Mydriasis (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1
Ocular icterus (Eye disorders) | 2 | 0
Ocular surface disease (Eye disorders) | 0 | 1
Panophthalmitis (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 5 | 5
Visual acuity reduced (Eye disorders) | 2 | 0
Vitreous floaters (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 30 | 24
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 15 | 22
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Aphagia (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 5 | 2
Aptyalism (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 5 | 2
Breath odour (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 4
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 29 | 42
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 335 | 188
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 11 | 15
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 41 | 34
Dysphagia (Gastrointestinal disorders) | 10 | 6
Enteritis (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 7 | 8
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 8 | 1
Gastritis atrophic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 6
Gingival bleeding (Gastrointestinal disorders) | 6 | 3
Gingivitis (Gastrointestinal disorders) | 3 | 0
Glossitis (Gastrointestinal disorders) | 1 | 1
Glossodynia (Gastrointestinal disorders) | 6 | 4
Haematemesis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 7 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 6 | 3
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 3 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Jejunitis (Gastrointestinal disorders) | 1 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 2 | 1
Lip oedema (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 2 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 114 | 90
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 3 | 3
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 5 | 6
Rectal haemorrhage (Gastrointestinal disorders) | 9 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 28 | 21
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1
Tongue haemorrhage (Gastrointestinal disorders) | 1 | 0
Tooth deposit (Gastrointestinal disorders) | 0 | 1
Tooth discolouration (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Tooth loss (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 3
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 86 | 66
Asthenia (General disorders) | 49 | 50
Axillary pain (General disorders) | 0 | 2
Catheter site pain (General disorders) | 1 | 1
Chest discomfort (General disorders) | 5 | 1
Chest pain (General disorders) | 44 | 47
Chills (General disorders) | 8 | 6
Condition aggravated (General disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 1
Discomfort (General disorders) | 1 | 0
Disease progression (General disorders) | 2 | 5
Face oedema (General disorders) | 2 | 0
Fatigue (General disorders) | 128 | 100
Feeling abnormal (General disorders) | 0 | 1
Feeling cold (General disorders) | 3 | 1
Gait disturbance (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 3 | 3
Hyperpyrexia (General disorders) | 3 | 0
Impaired healing (General disorders) | 0 | 1
Implant site discharge (General disorders) | 1 | 0
Influenza like illness (General disorders) | 5 | 2
Malaise (General disorders) | 2 | 2
Medical device complication (General disorders) | 1 | 0
Mucosal dryness (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 40 | 27
Mucous membrane disorder (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 0
Oedema (General disorders) | 4 | 6
Oedema peripheral (General disorders) | 27 | 26
Pain (General disorders) | 4 | 10
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 43 | 37
Sensation of foreign body (General disorders) | 0 | 1
Ulcer (General disorders) | 0 | 1
Vestibulitis (General disorders) | 0 | 1
Xerosis (General disorders) | 2 | 1
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 1 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 23 | 6
Jaundice (Hepatobiliary disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal wall infection (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 2 | 0
Abscess limb (Infections and infestations) | 2 | 1
Abscess oral (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Anal fungal infection (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 12 | 14
Bronchopneumonia (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 4 | 4
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 9 | 5
Dermatitis infected (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 1 | 2
Erysipelas (Infections and infestations) | 2 | 0
Eye infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 6 | 7
Fungal infection (Infections and infestations) | 0 | 2
Fungal skin infection (Infections and infestations) | 0 | 7
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3
H1N1 influenza (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 3
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 4 | 4
Influenza (Infections and infestations) | 7 | 13
Labyrinthitis (Infections and infestations) | 2 | 1
Localised infection (Infections and infestations) | 7 | 3
Lower respiratory tract infection (Infections and infestations) | 9 | 10
Lung infection (Infections and infestations) | 1 | 3
Lymphangitis (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 9 | 14
Onychomycosis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 9 | 3
Oral fungal infection (Infections and infestations) | 1 | 5
Oral herpes (Infections and infestations) | 2 | 0
Oral infection (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 2
Otitis media (Infections and infestations) | 1 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 25 | 19
Pharyngitis (Infections and infestations) | 5 | 4
Pneumonia (Infections and infestations) | 14 | 17
Pulpitis dental (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 5 | 3
Respiratory tract infection (Infections and infestations) | 7 | 6
Rhinitis (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 2
Skin bacterial infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 3
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 3
Tonsillitis (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 2 | 0
Tracheitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 12
Urinary tract infection (Infections and infestations) | 13 | 15
Vaginal infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 1 | 2
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Inappropriate schedule of drug administration (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 2 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 13 | 11
Aspartate aminotransferase increased (Investigations) | 12 | 10
Aspiration bronchial (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 10
Blood bilirubin increased (Investigations) | 3 | 1
Blood calcium increased (Investigations) | 1 | 1
Blood creatine increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 6 | 4
Blood lactate dehydrogenase increased (Investigations) | 6 | 5
Blood magnesium decreased (Investigations) | 2 | 0
Blood phosphorus decreased (Investigations) | 1 | 1
Blood potassium decreased (Investigations) | 2 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 4 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 2
Blood urea decreased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 2 | 2
Blood uric acid decreased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 2
Body temperature decreased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 2 | 2
Breath sounds abnormal (Investigations) | 4 | 5
C-reactive protein increased (Investigations) | 4 | 2
Cardiac murmur (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 1
Eastern cooperative oncology group performance status worsened (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 2
Fibrin D dimer increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 7 | 8
Heart rate irregular (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hypophonesis (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 6 | 3
Platelet count increased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 1 | 1
Renal function test abnormal (Investigations) | 0 | 1
Thrombin time prolonged (Investigations) | 0 | 1
Thyroxine increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 79 | 64
Weight increased (Investigations) | 3 | 0
White blood cell count decreased (Investigations) | 4 | 0
White blood cell count increased (Investigations) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 190 | 133
Dehydration (Metabolism and nutrition disorders) | 13 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3
Fluid retention (Metabolism and nutrition disorders) | 2 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 33 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 6
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 4
Malnutrition (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 17
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 32
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 14
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 19
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 13
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 9
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 14
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 26
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Palmar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Acrodynia (Nervous system disorders) | 1 | 0
Ageusia (Nervous system disorders) | 10 | 1
Anosmia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Areflexia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 2
Burning sensation (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Clonus (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 21 | 27
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 64 | 27
Dyslalia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 1
Facial neuralgia (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Facial spasm (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 25 | 23
Horner's syndrome (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypertonia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 4
Hypogeusia (Nervous system disorders) | 3 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 4 | 4
Memory impairment (Nervous system disorders) | 1 | 1
Monoplegia (Nervous system disorders) | 1 | 1
Motor dysfunction (Nervous system disorders) | 1 | 1
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 6 | 5
Paraesthesia (Nervous system disorders) | 7 | 8
Peripheral motor neuropathy (Nervous system disorders) | 3 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 9
Petit mal epilepsy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 6
Presyncope (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 6 | 2
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 4
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 4 | 3
Vagus nerve disorder (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 19 | 17
Confusional state (Psychiatric disorders) | 6 | 3
Delirium (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 15 | 15
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 21 | 28
Listless (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 2 | 1
Nervousness (Psychiatric disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 3
Sopor (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Albuminuria (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Choluria (Renal and urinary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 9 | 7
Haematuria (Renal and urinary disorders) | 7 | 4
Haemoglobinuria (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 21 | 10
Renal colic (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 2 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 2
Urine flow decreased (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast discharge (Reproductive system and breast disorders) | 0 | 1
Breast oedema (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Genital rash (Reproductive system and breast disorders) | 2 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 4
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 81 | 96
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 13 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 95 | 103
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 43 | 21
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 34 | 29
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 9 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 18
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 65 | 64
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 52 | 58
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 12
Exfoliative rash (Skin and subcutaneous tissue disorders) | 4 | 6
Hair colour changes (Skin and subcutaneous tissue disorders) | 8 | 2
Hair disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 3
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 2 | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discomfort (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 8
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 42 | 20
Periorbital oedema (Skin and subcutaneous tissue disorders) | 2 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 5 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 53
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 277 | 255
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 2
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 5 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 13
Rash papular (Skin and subcutaneous tissue disorders) | 6 | 6
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 3
Rash scarlatiniform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 3 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 5 | 14
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin maceration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 5 | 0
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 7 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Urethral dilation procedure (Surgical and medical procedures) | 0 | 1
Angiodysplasia (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Flushing (Vascular disorders) | 2 | 2
Haematoma (Vascular disorders) | 3 | 1
Hot flush (Vascular disorders) | 5 | 1
Hyperaemia (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 37 | 11
Hypotension (Vascular disorders) | 5 | 5
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0
Pallor (Vascular disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 2 | 1
Phlebitis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 1 | 3
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 2
Venous insufficiency (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.